CLINICAL TRIAL: NCT03141996
Title: Use of Vibration to Improve Visual/Spatial Neglect in Patients Affected by Stroke
Acronym: NEGLECT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NEGLECT STUDY
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Unilateral Spatial Neglect
Keywords: vibration; stroke; activities of daily living
MeSH Terms: conditions — Stroke | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vibration to upper posterior neck muscles (Experimental): Treatment will be performed by occupational therapist practitioners prior to regular occupational therapy session using a vibration tool.
  Interventions: Other: Vibration to upper posterior neck muscles
- Standard of care (Active Comparator): Regular occupational therapy session
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Vibration to upper posterior neck muscles — Vibration to upper posterior neck muscles using a vibrational tool.
  Other Names: Magic Wand Massager
  Arms: Vibration to upper posterior neck muscles
Other: Standard of Care — Standard of care treatment
  Arms: Standard of care

SUMMARY:
This study will measure if five minutes of vibration to the upper back neck muscles, prior to standard of care treatment, will improve symptoms of spatial neglect and/or activities of daily living function for patients who have had a stroke.

DETAILED DESCRIPTION:
Spatial neglect is a common syndrome following stroke, most frequently of the right side of the brain. Such patients fail to be aware of objects or people to their left. This study is being done to learn if vibration treatment can improve visual/spatial neglect and activities of daily living in stroke patients better than current standard intervention.This treatment will be performed by occupational therapist practitioners prior to regular occupational therapy session using a vibration tool.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* demonstrated visual/spatial neglect, as demonstrated by NIH Stroke Scale (NIHSS) and deficits in assessing tactile extinction and visuospatial neglect done on admission.

Exclusion Criteria:

* severe pain or skin disease at the posterior neck
* severe atherosclerosis of carotid arteries by an ultrasonic evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-04-16 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-04-12 (Actual)

PRIMARY OUTCOMES:
Behavioral Inattention test | Day 0
  A short screening battery of tests to assess the presence and the extent of visual neglect on a sample of everyday problems faced by patients

SECONDARY OUTCOMES:
Behavioral Inattention test | Day 30
  A short screening battery of tests to assess the presence and the extent of visual neglect on a sample of everyday problems faced by patients
Behavioral Inattention test | Day 60
  A short screening battery of tests to assess the presence and the extent of visual neglect on a sample of everyday problems faced by patients
Catherine Bergego Scale (CBS) | Day 0
  a standardized checklist to detect presence and degree of unilateral neglect during observation of everyday life situations.
Catherine Bergego Scale (CBS) | Day 30
  a standardized checklist to detect presence and degree of unilateral neglect during observation of everyday life situations.
Catherine Bergego Scale (CBS) | Day 90
  a standardized checklist to detect presence and degree of unilateral neglect during observation of everyday life situations.
Activity Measure for Post-Acute Care (AM-PAC) | Day 0
  AM-PAC measures patients' capabilities in functional areas for prioritization of therapy resources.
Activity Measure for Post-Acute Care (AM-PAC) | Day 30
  AM-PAC measures patients' capabilities in functional areas for prioritization of therapy resources.
Activity Measure for Post-Acute Care (AM-PAC) | Day 60
  AM-PAC measures patients' capabilities in functional areas for prioritization of therapy resources.

CONTACTS AND LOCATIONS:
Overall Officials: Florentina Mueller-Planitz, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Longley V, Hazelton C, Heal C, Pollock A, Woodward-Nutt K, Mitchell C, Pobric G, Vail A, Bowen A. Non-pharmacological interventions for spatial neglect or inattention following stroke and other non-progressive brain injury. Cochrane Database Syst Rev. 2021 Jul 1;7(7):CD003586. doi: 10.1002/14651858.CD003586.pub4. PMID 34196963